CLINICAL TRIAL: NCT05467865
Title: A Quasi-experimental Intervention Protocol for Nutrition Education About Celiac Disease to Primary School Children (Zeliakide Project)
Brief Title: Celiac Disease: Nutrition Education in Primary School
Acronym: ZELIAKIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, Itziar Churruca Ortega, Profesor Titular de Universidad - University Tenured Professor, University of the Basque Country (UPV/EHU)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: M10_2020_081 ZELIAKIDE; GIU18/078 (Other Grant/Funding Number: Basque Government); IT1419-19 (Other Grant/Funding Number: University of the Basque Country (UPV/EHU))
Record Dates: First submitted 2022-04-26; First posted 2022-07-21 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Celiac Disease
Keywords: celiac disease; nutrition education; children; gluten-free diet; balanced diet
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental, nutrition education program (Experimental)
  Interventions: Other: ZELIAKIDE
- control group (No Intervention)

INTERVENTIONS:
Other: ZELIAKIDE — The nutrition education program will be adapted to the curriculum of the schools. The intervention will consist of 8 sessions and the main topics will be: (1) to understand the balanced diet and to apply it to one´s own diet, (2) to learn what celiac disease and gluten are, (3) to promote social inclusion.
  Each session will last 60 minutes and they will take place during school hours. The whole intervention will last 4 weeks, 2 sessions per week. Teaching-learning process will be developed through games and experiments.
  Designed activities are based on IBL methodology, which has proven to be very effective in science teaching-learning processes. As a result, inquiry-oriented TLS has been developed, focused on facilitating children's understanding of the research process.
  Arms: Experimental, nutrition education program

SUMMARY:
Celiac disease is a chronic immune-based intestinal pathology. Its prevalence is 1% and its incidence has increased in recent years. This disease usually causes gastrointestinal and/or extraintestinal symptoms, which can only be reduced by following a strict, lifelong gluten-free diet. In addition, the social life of people with celiac disease is impaired due to the impact of the gluten-free diet on daily activities.

An adequate Nutrition Education program can improve the physical and social health of these people. Moreover, considering the high impact this disease has on the people close to the celiac patient, and due to the important role that general population has in the care and inclusion of persons with celiac disease, education should be directed to general population.

Therefore, the purpose of ZELIAKIDE program is to promote Nutrition Education in general population. In particular, the specific aims are 1) to promote the social inclusion of people with celiac disease by raising awareness among the general population, and 2) to promote a balanced diet and an interest in science and research among children.

ZELIAKIDE is an intervention aimed at children and focused on the school environment, and is based on Inquiry Based Learning (IBL) methodology. Inquiry-based Teaching-Learning Sequence (TLS) has been created to internalize and integrate competences related to celiac disease, gluten, gluten-free diet, balanced diet and healthy lifestyle.

In addition, this TLS aims to develop scientific competence through activities that promote science and the research process.

Although nutrition education programs for children have proven to be effective, it has been observed that children's interest in science has decreased. The investigators therefore aim to implement a nutrition education programme based on previous experiences that promotes science skills and stimulates children's interest in science.

ELIGIBILITY:
Inclusion Criteria:

* School must show interest in participating in the project.
* Children study in a primary school that must be used to project based learning.
* Have at least one class in grades 5th and 6th level of primary school.

Exclusion Criteria:

* Family or closed relationship with school students.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 299 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Change in nutrition knowledge | 4 weeks, twice a week
  A questionnaire was designed to be able to assess all outcomes. It was divided into 8 parts: each one for each session, carried out in different days. The same questionnaire part is completed twice (before and after each session) in order to assess changes due to the intervention.
  Regarding the change in nutrition knowledge will be measured in parts 1 and 2 of the questionnaire. The unit of measure will be the score obtained in the questionnaires (0, worst - 4, best / the number of correct answers).
Change in Celiac Disease knowledge | 4 weeks, twice a week
  The questionnaire will be used to measure the change (see explanation of the type of questionnaire in the first outcome measure). The change in Celiac Disease knowledge will be measured in part 3 of the questionnaire. The unit of measure will be the score obtained in the questionnaires (0, worst - 4, best / the number of correct answers).
Change in intentional behavior related to the social inclusion of people with Celiac condition | 4 weeks, twice a week
  The questionnaire will be used to measure the change (see explanation of the type of questionnaire in the first outcome measure). The change in intentional behavior will be measured in part 3, 6 and 8 of the questionnaire. The unit of measure will be the score obtained in the questionnaires (0, worst - 4, best / the number of correct answers).
Change in knowledge regarding gluten and its presence in food | 4 weeks, twice a week
  The questionnaire will be used to measure the change (see explanation of the type of questionnaire in the first outcome measure). The change in knowledge regarding gluten and its presence in food will be measured in part 3, 4, 5, and 7 of the questionnaire. The unit of measure will be the score obtained in the questionnaires (0, worst - 4, best / the number of correct answers).
Change in behavior in relation to interest in science | 4 weeks, twice a week
  The questionnaire will be used to measure the change (see explanation of the type of questionnaire in the first outcome measure). The change in knowledge regarding gluten and its presence in food will be measured in part 5 of the questionnaire. The unit of measure will be the score obtained in the questionnaires in order to assess behavior change (0, worst; 4, best).
Change in behavior in relation to the consumption of unhealthy foods | 4 weeks, twice a week
  The questionnaire will be used to measure the change in behavior in relation to the consumption of unhealthy foods, it will be measured in parts 2-8. The unit of measure will be the score obtained in the questionnaires (0, worst - 5, best).

SECONDARY OUTCOMES:
Opinion of the parents/guardians of the children in relation to the project | immediately after the intervention.
  A separate questionnaire will be completed by parents/guardians of the participants. This questionnaire will measure the two secondary outcomes. The answers to the questionnaire will be yes/no/don't know.
Opinion of the children about the project reported by their parents/guardians | immediately after the intervention.
  A separate questionnaire will be completed by parents/guardians of the participants. This questionnaire will measure the two secondary outcomes. The answers to the questionnaire will be yes/no/don't know.

CONTACTS AND LOCATIONS:
Locations (1):
- Itziar Churruca Ortega, Vitoria-Gasteiz, Álava, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sevinc E, Cetin FH, Coskun BD. Psychopathology, quality of life, and related factors in children with celiac disease. J Pediatr (Rio J). 2017 May-Jun;93(3):267-273. doi: 10.1016/j.jped.2016.06.012. Epub 2016 Nov 23. PMID 27886806
- [Background] Murimi MW, Kanyi M, Mupfudze T, Amin MR, Mbogori T, Aldubayan K. Factors Influencing Efficacy of Nutrition Education Interventions: A Systematic Review. J Nutr Educ Behav. 2017 Feb;49(2):142-165.e1. doi: 10.1016/j.jneb.2016.09.003. Epub 2016 Nov 1. PMID 27814976
- [Background] Lasa A, Larretxi I, Simon E, Churruca I, Navarro V, Martinez O, Bustamante MA, Miranda J. New Software for Gluten-Free Diet Evaluation and Nutritional Education. Nutrients. 2019 Oct 17;11(10):2505. doi: 10.3390/nu11102505. PMID 31627463
- [Background] Haas K, Martin A, Park KT. Text Message Intervention (TEACH) Improves Quality of Life and Patient Activation in Celiac Disease: A Randomized Clinical Trial. J Pediatr. 2017 Jun;185:62-67.e2. doi: 10.1016/j.jpeds.2017.02.062. Epub 2017 Mar 23. PMID 28343658
- [Background] Halmos EP, Deng M, Knowles SR, Sainsbury K, Mullan B, Tye-Din JA. Food knowledge and psychological state predict adherence to a gluten-free diet in a survey of 5310 Australians and New Zealanders with coeliac disease. Aliment Pharmacol Ther. 2018 Jul;48(1):78-86. doi: 10.1111/apt.14791. Epub 2018 May 7. PMID 29733115
- [Background] Patriota PF, Filgueiras AR, de Almeida VBP, Alexmovitz GAC, da Silva CE, de Carvalho VFF, Carvalho N, de Albuquerque MP, Domene SMA, do Prado WL, Torres GES, de Oliveira APR, Sesso R, Sawaya AL. Effectiveness of a 16-month multi-component and environmental school-based intervention for recovery of poor income overweight/obese children and adolescents: study protocol of the health multipliers program. BMC Public Health. 2017 Sep 15;17(1):708. doi: 10.1186/s12889-017-4715-8. PMID 28915797
- [Background] Li B, Pallan M, Liu WJ, Hemming K, Frew E, Lin R, Liu W, Martin J, Zanganeh M, Hurley K, Cheng KK, Adab P. The CHIRPY DRAGON intervention in preventing obesity in Chinese primary-school--aged children: A cluster-randomised controlled trial. PLoS Med. 2019 Nov 26;16(11):e1002971. doi: 10.1371/journal.pmed.1002971. eCollection 2019 Nov. PMID 31770371
- [Background] Minossi V, Pellanda LC. The "Happy Heart" educational program for changes in health habits in children and their families: protocol for a randomized clinical trial. BMC Pediatr. 2015 Mar 10;15:19. doi: 10.1186/s12887-015-0336-5. PMID 25885095
- [Background] Gold A, Larson M, Tucker J, Strang M. Classroom Nutrition Education Combined With Fruit and Vegetable Taste Testing Improves Children's Dietary Intake. J Sch Health. 2017 Feb;87(2):106-113. doi: 10.1111/josh.12478. PMID 28076921
- [Background] Wall DE, Least C, Gromis J, Lohse B. Nutrition education intervention improves vegetable-related attitude, self-efficacy, preference, and knowledge of fourth-grade students. J Sch Health. 2012 Jan;82(1):37-43. doi: 10.1111/j.1746-1561.2011.00665.x. PMID 22142173
- [Derived] Vazquez-Polo M, Churruca I, Lasa A, Perez-Junkera G, Larretxi I, Bustamante MA, Martinez O, Navarro V. Effectiveness of a controlled trial of nutrition education in primary school, ZELIAKIDE project: knowledge and mid-morning snack consumption. BMC Public Health. 2025 Dec 23. doi: 10.1186/s12889-025-25821-3. Online ahead of print. PMID 41437238